CLINICAL TRIAL: NCT03277833
Title: Efficacy and Safety of Gynostemma Pentaphyllum(Dungkulcha) Extract on Alleviation of Chronic Stress-induced Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CBU-STR-DOLWOE
Record Dates: First submitted 2016-05-13; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Chronic Stress-Induced Strain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gynostemma Pentaphyllum(Dungkulcha) Extract (Experimental): Gynostemma Pentaphyllum(Dungkulcha) Extract (400mg/d)
  Interventions: Dietary Supplement: Gynostemma Pentaphyllum(Dungkulcha) Extract(400mg/day)
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gynostemma Pentaphyllum(Dungkulcha) Extract(400mg/day) — Gynostemma Pentaphyllum(Dungkulcha) Extract(400mg/day), parallel design
  Arms: Gynostemma Pentaphyllum(Dungkulcha) Extract
Dietary Supplement: Placebo — Placebo, parallel design
  Arms: Placebo

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Gynostemma Pentaphyllum(Dungkulcha) on alleviation of chronic stress-induced strain. The investigators measured decrement of body fat parameters, State&Trait version of STAI, Beck Anxiety Inventory(BAI), Hamilton Anxiety Inventory(HAM-A), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

• Age 20-65 years with chronic stress( S-STAI score 40~60)

Exclusion Criteria:

* excessive physically chronic fatigue
* Subjects taking antidepressants, anxiolytics, hypnotics within the last 2 months prior to the study
* Cardiovascular disease
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Renal disease
* Abnormal hepatic function
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* History of alcohol or substance abuse
* Pregnancy or lacting women etc.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in score of State&Trait version of STAI | Baseline and 8 weeks
  Score of State&Trait version of STAI was measured in study screening and visit 3(8 week).

SECONDARY OUTCOMES:
Change of Blood Norepinephrine Level | Baseline and 8 week
  Blood norepinephrine level was measured in study visit 1(0 week) and visit 3(8 week).
Change of Blood Cortisol Level | Baseline and 8 week
  Blood cortisol level was measured in study visit 1(0 week) and visit 3(8 week).
Change in score of Beck Anxiety Inventory | Baseline and 8 week
  Score of Beck Anxiety Inventory was measured in study visit 1(0 week) and visit 3(8 week).

IPD SHARING:
Plan to Share IPD: No